CLINICAL TRIAL: NCT03486392
Title: A Randomized, Double-blind Placebo-controlled and Open-label Active-controlled, Parallel-group, Multicenter, Dose-ranging Study to Evaluate the Safety and Efficacy of JNJ-64565111 in Non-diabetic Severely Obese Subjects
Brief Title: A Study to Evaluate the Safety and Efficacy of JNJ-64565111 in Non-diabetic Severely Obese Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108314; 64565111OBE2001 (Other: Janssen Research & Development, LLC); 2017-003616-39 (EudraCT Number)
Record Dates: First submitted 2018-03-23; First posted 2018-04-03 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Double-Blind: JNJ-64565111 Dose Level 1 (Experimental): Participants will receive a JNJ-64565111 Dose Level 1 subcutaneously (SC) once-weekly for 26-week treatment phase.
  Interventions: Drug: JNJ-64565111 Dose Level 1
- Double-Blind: JNJ-64565111 Dose Level 2 (Experimental): Participants will receive a JNJ-64565111 Dose Level 2 SC once-weekly for 26-week treatment phase.
  Interventions: Drug: JNJ-64565111 Dose Level 2
- Double-Blind: JNJ-64565111 Dose Level 3 (Experimental): Participants will receive a JNJ-64565111 Dose Level 3 SC once-weekly for 26-week treatment phase.
  Interventions: Drug: JNJ-64565111 Dose Level 3
- Double-Blind: Placebo (Placebo Comparator): Participants will receive placebo matching to JNJ-64565111 SC once-weekly for 26-week treatment phase.
  Interventions: Drug: Placebo
- Open-Label: 3.0 milligram (mg) Liraglutide (Active Comparator): Participant will receive once-daily doses of 0.6, 1.2, 1.8, 2.4, or 3.0 mg. The participants will receive liraglutide at a starting dose of 0.6 mg SC once-daily on Day 1. Participants will be instructed to increase the dose of liraglutide by 0.6 mg dose increment every 7 days, up to the full dosage of 3.0 mg by Week 5. Participants will then continue on the 3.0 mg once-daily dosage until Week 26.
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: JNJ-64565111 Dose Level 1 — Participants will receive JNJ-64565111 Dose Level 1 SC once -weekly until Week 26.
  Arms: Double-Blind: JNJ-64565111 Dose Level 1
Drug: JNJ-64565111 Dose Level 2 — Participants will receive JNJ-64565111 Dose Level 2 SC once-weekly until Week 26.
  Arms: Double-Blind: JNJ-64565111 Dose Level 2
Drug: JNJ-64565111 Dose Level 3 — Participants will receive JNJ-64565111 Dose Level 3 SC once-weekly until Week 26.
  Arms: Double-Blind: JNJ-64565111 Dose Level 3
Drug: Liraglutide — Participants will receive liraglutide at a starting dose of 0.6 mg then dose will be ramped up by 0.6 mg daily until reaching 3.0 mg. Participants will then continue on the 3.0 mg once-daily dosage until Week 26.
  Other Names: Saxenda
  Arms: Open-Label: 3.0 milligram (mg) Liraglutide
Drug: Placebo — Participants will receive matching placebo SC once-weekly until Week 26.
  Arms: Double-Blind: Placebo

SUMMARY:
The purpose of this study is to assess the effects of JNJ-64565111 compared with placebo after 26 weeks of treatment on the percent change in body weight from baseline and to assess the safety and tolerability, in non-diabetic severely obese participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) greater than or equal to (>=) 35 to less than or equal to (<=) 50 kilogram per square meter (kg/m^2) at the screening visit
* Stable weight (that is, change of <= 5 percent [%] within 12 weeks before screening based on medical history)
* Women must be either: (a) Postmenopausal, or (b) Permanently sterilized or otherwise be incapable of pregnancy, or (c) Heterosexually active and practicing a highly effective method of birth control, or (d) Not heterosexually active
* Woman of childbearing potential have a negative pregnancy test at screening
* Willing and able to adhere to specific the prohibitions and restrictions

Exclusion Criteria:

* History of obesity with a known secondary cause (for example, Cushing's disease/syndrome)
* History of Type 1 diabetes mellitus, Type 2 diabetes mellitus (T2DM), diabetic ketoacidosis (DKA), pancreas or beta-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy
* Has a Hemoglobin A1c (HbA1c) of >= 6.5% or fasting plasma glucose (FPG) >= 126 milligrams per deciliter (mg/dL) (>= 7.0 millimoles per liter [mmol/L]) at screening
* Screening calcitonin of >= 50 picograms per milliliter (pg/mL) personal history or family history of medullary thyroid cancer, or of multiple endocrine neoplasia syndrome type 2 (MEN 2), regardless of time prior to screening
* History of glucagonoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (51):
- United States (17):
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Care Partners Clinical Research, Jacksonville, Florida
  - Advanced Clinical Research, Boise, Idaho
  - Medisphere Medical Research Center, Llc, Evansville, Indiana
  - L-Marc Research Center, Louisville, Kentucky
  - Milford Emergency Associates, Inc., Marlborough, Massachusetts
  - Central New York Clinical Research, Manlius, New York
  - Weill Cornell Medicine, New York, New York
  - Rapid Medical Research, Cleveland, Ohio
  - Omega Medical Research, Warwick, Rhode Island
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Dallas Diabetes Research Center, Dallas, Texas
  - Permian Research Foundation, Odessa, Texas
  - Advanced Clinical Research, West Jordan, Utah
  - Rainier Clinical Research Center, Renton, Washington
  - Allegiance Reserach Specialists, LLC, Wauwatosa, Wisconsin
- Belgium (8):
  - OLV Ziekenhuis Aalst, Aalst
  - CSL Arlon, Arlon
  - UZ Antwerpen, Edegem
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
  - AZ Delta, Roeselare
  - AZ Glorieux Ronse, Ronse
  - Practimed Medical Center, Tessenderlo
- Canada (7):
  - Joanne F. Liutkus Medicine Professional Corporation, Cambridge, Ontario
  - Canadian Phase Onward, Toronto, Ontario
  - Dr. Anil K Gupta Medicine Professional Corporation, Toronto, Ontario
  - Manna Research, Toronto, Ontario
  - Manna Research, Lévis, Quebec
  - Manna Research, Pointe-Claire, Quebec
  - Clinique des Maladies Lipidiques de Québec, Québec, Quebec
- Poland (5):
  - Indywidualna Praktyka Lekarska, Gabinet Leczenia Otyłości i Chorób Dietozależnych, Bialystok
  - Centrum Badań Klinicznych PI-House sp. z o.o., Gdansk
  - NZOZ 'Linia' Centrum Leczenia Zaburzeń Metabolicznych Magdalena Olszanecka-Glinianowicz, Katowice
  - Nzoz Salvia, Katowice-Ligota
  - Centrum Zdrowia Metabolicznego Paweł Bogdański, Poznan
- Sweden (7):
  - Katarina Berndtsson-Blom Ladulaaskliniken, Borås
  - Intern Medicin, Gothenburg
  - PTC,Primary care Trial Center, Gothenburg
  - PharmaSite, Helsingborg
  - PharmaSite, Malmo
  - Avdelningen för kliniska prövningar, Örebro
  - PTC- Skaraborg, Skövde
- United Kingdom (7):
  - Southmead Hospital, Bristol
  - Ashgate Medical Practice, Chesterfield
  - Hathaway Medical Centre, Chippenham
  - Aintree University Hospital NHS Trust, Liverpool
  - Clifton Medical Centre, Rotherham
  - Albany House Medical Centre, Wellingborough
  - Bradford on Avon and Melksham Health Partnership, Wiltshire

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 474 participants were randomized out of which 444 participants completed the study.
Groups:
- Double Blind: Placebo: Participants self-administered the matching placebo of JNJ-64565111 subcutaneously (SC) once-weekly throughout the 26-week treatment phase or until early discontinuation of study drug.
- Double Blind: JNJ-64565111 5.0 mg: Participants self-administered 5.0 milligram (mg) JNJ-64565111 SC once weekly throughout the 26-week treatment phase or until early discontinuation of study drug.
- Double Blind: JNJ-64565111 7.4 mg: Participants self-administered 7.4 mg JNJ-64565111 SC once-weekly throughout the 26-week treatment phase or until early discontinuation of study drug.
- Double Blind: JNJ-64565111 10.0 mg: Participants self-administered 10.0 mg JNJ-64565111 SC once-weekly throughout the 26-week treatment phase or until early discontinuation of study drug.
- Open Label: Liraglutide 3.0 mg: Participant self-administered liraglutide at a starting dose of 0.6 mg SC once-daily on Day 1, followed by dose titration up to 1.2, 1.8, 2.4, and 3.0 mg in Weeks 2, 3, 4, and 5 (with 0.6 mg weekly increment up to the full dosage of 3.0 mg by Week 5). Participants then continued the 3.0 mg once-daily dosage until Week 26 or until early drug discontinuation.
Period: Overall Study
Arm/Group | Double Blind: Placebo | Double Blind: JNJ-64565111 5.0 mg | Double Blind: JNJ-64565111 7.4 mg | Double Blind: JNJ-64565111 10.0 mg | Open Label: Liraglutide 3.0 mg
Started | 60 | 59 | 118 | 118 | 119
Completed | 57 | 59 | 104 | 109 | 115
Not Completed | 3 | 0 | 14 | 9 | 4
Not completed — Lost to Follow-up | 0 | 0 | 8 | 5 | 2
Not completed — Withdrawal by Subject | 3 | 0 | 6 | 4 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double Blind: Placebo | Double Blind: JNJ-64565111 5.0 mg | Double Blind: JNJ-64565111 7.4 mg | Double Blind: JNJ-64565111 10.0 mg | Open Label: Liraglutide 3.0 mg | Total
Number analyzed (Participants) | 60 | 59 | 118 | 118 | 119 | 474
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (11.84) | 47.3 (11.18) | 46.2 (11.68) | 46.2 (12.16) | 45.6 (11.71) | 46.3 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 47 | 86 | 86 | 89 | 356
  Male | 12 | 12 | 32 | 32 | 30 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 9 | 11 | 14 | 42
  Not Hispanic or Latino | 57 | 54 | 108 | 107 | 105 | 431
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 1 | 1 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 3 | 1 | 4
  Black or African American | 8 | 3 | 8 | 8 | 7 | 34
  White | 51 | 56 | 106 | 103 | 105 | 421
  More than one race | 0 | 0 | 2 | 2 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 7 | 5 | 15 | 13 | 18 | 58
  CANADA | 9 | 8 | 12 | 17 | 16 | 62
  POLAND | 8 | 6 | 14 | 18 | 15 | 61
  SWEDEN | 12 | 14 | 22 | 19 | 14 | 81
  UNITED KINGDOM | 5 | 8 | 17 | 11 | 17 | 58
  UNITED STATES | 19 | 18 | 38 | 40 | 39 | 154

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Body Weight at Week 26
Description: Percent change in body weight in kilograms (kg) from baseline to Week 26 was reported.
Time Frame: Baseline, Week 26
Population: Modified intent-to-treat (mITT) population included all ITT participants who had taken at least 1 dose of study drug and had at least 1 post-baseline body weight measurement; for liraglutide, only those who titrated to 3.0 mg were included in mITT population. N (number of participants analyzed) = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Groups:
- Double Blind: JNJ-64565111 5.0 mg: Participants self-administered 5.0 milligram (mg) JNJ-64565111 SC once-weekly throughout the 26-week treatment phase or until early discontinuation of study drug.
Arm/Group | Double Blind: Placebo | Double Blind: JNJ-64565111 5.0 mg | Double Blind: JNJ-64565111 7.4 mg | Double Blind: JNJ-64565111 10.0 mg | Open Label: Liraglutide 3.0 mg
Number analyzed (Participants) | 60 | 58 | 109 | 109 | 108
Percent Change | -1.76 (0.73) | -8.51 (0.76) | -9.83 (0.56) | -11.80 (0.58) | -7.54 (0.54)
Statistical Analysis 1: Comparison: Double Blind: Placebo vs Double Blind: JNJ-64565111 5.0 mg; Test type: Superiority; p < 0.001, Dunnett's method; Difference of least square (LS) Means = -6.75, 95% CI 2-sided [-9.31 to -4.19], Standard Error of Mean 1.056
Statistical Analysis 2: Comparison: Double Blind: Placebo vs Double Blind: JNJ-64565111 7.4 mg; Test type: Superiority; p < 0.001, Dunnett's method; Difference of LS Means = -8.07, 95% CI 2-sided [-10.31 to -5.84], Standard Error of Mean 0.921
Statistical Analysis 3: Comparison: Double Blind: Placebo vs Double Blind: JNJ-64565111 10.0 mg; Test type: Superiority; p < 0.001, Dunnett's method; Difference of LS Means = -10.04, 95% CI 2-sided [-12.31 to -7.78], Standard Error of Mean 0.934
Statistical Analysis 4: Comparison: Double Blind: Placebo vs Open Label: Liraglutide 3.0 mg; Test type: Superiority; p < 0.001, Dunnett's method; Difference of LS Means = -5.78, 95% CI 2-sided [-7.99 to -3.57], Standard Error of Mean 0.910

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. A TEAE was defined as an AE with an onset after the initiation study drug and before the last study drug date of the double-blind (26-week) treatment phase for plus 28 days for liraglutide participants, and plus 35 days for JNJ-64565111 and placebo participants.
Time Frame: Up to Week 30
Population: Safety analysis set included all randomized participants who had received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind: Placebo | Double Blind: JNJ-64565111 5.0 mg | Double Blind: JNJ-64565111 7.4 mg | Double Blind: JNJ-64565111 10.0 mg | Open Label: Liraglutide 3.0 mg
Number analyzed (Participants) | 60 | 59 | 118 | 118 | 119
Participants | 43 | 53 | 110 | 110 | 96

3. Secondary Outcome: Number of Participants With Greater Than or Equal to (>=) 5 Percent (%) Body Weight Loss at Week 26
Description: Number of participants with >= 5% body weight loss from baseline to Week 26 were reported.
Time Frame: Week 26
Population: mITT population included all ITT participants who had taken at least 1 dose of study drug and had at least 1 post-baseline body weight measurement; for liraglutide, only those who titrated to 3.0 mg were included in mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind: Placebo | Double Blind: JNJ-64565111 5.0 mg | Double Blind: JNJ-64565111 7.4 mg | Double Blind: JNJ-64565111 10.0 mg | Open Label: Liraglutide 3.0 mg
Number analyzed (Participants) | 60 | 59 | 116 | 116 | 109
Participants | 8 | 34 | 70 | 62 | 56

4. Secondary Outcome: Number of Participants With Greater Than or Equal to 10 % Body Weight Loss at Week 26
Description: Number of participants with >= 10 % body weight loss from baseline to Week 26 were reported.
Time Frame: Week 26
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind: Placebo | Double Blind: JNJ-64565111 5.0 mg | Double Blind: JNJ-64565111 7.4 mg | Double Blind: JNJ-64565111 10.0 mg | Open Label: Liraglutide 3.0 mg
Number analyzed (Participants) | 60 | 59 | 116 | 116 | 109
Participants | 2 | 23 | 43 | 46 | 27

5. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: Change from baseline in body weight at Week 26 was reported.
Time Frame: Baseline, Week 26
Population: mITT population included all ITT participants who had taken at least 1 dose of study drug and had at least 1 post-baseline body weight measurement; for liraglutide, only those who titrated to 3.0 mg were included in mITT population. N (number of participants analyzed) = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Double Blind: Placebo | Double Blind: JNJ-64565111 5.0 mg | Double Blind: JNJ-64565111 7.4 mg | Double Blind: JNJ-64565111 10.0 mg | Open Label: Liraglutide 3.0 mg
Number analyzed (Participants) | 60 | 58 | 109 | 109 | 108
kg | -2.05 (0.827) | -9.58 (0.861) | -11.07 (0.633) | -13.23 (0.656) | -8.32 (0.610)

ADVERSE EVENTS:
Time Frame: Up to 30 Weeks
Description: Safety analysis set included all randomized participants who had received at least one dose of study drug.
Arm/Group | Double Blind: Placebo | Double Blind: JNJ-64565111 5.0 mg | Double Blind: JNJ-64565111 7.4 mg | Double Blind: JNJ-64565111 10.0 mg | Open Label: Liraglutide 3.0 mg
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/59 | 0/118 | 0/118 | 1/119
Serious Adverse Events (participants affected / at risk) | 4/60 | 3/59 | 2/118 | 4/118 | 4/119
Other Adverse Events (participants affected / at risk) | 33/60 | 43/59 | 106/118 | 104/118 | 81/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind: Placebo (N=60) | Double Blind: JNJ-64565111 5.0 mg (N=59) | Double Blind: JNJ-64565111 7.4 mg (N=118) | Double Blind: JNJ-64565111 10.0 mg (N=118) | Open Label: Liraglutide 3.0 mg (N=119)
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Stress Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Biliary Colic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Major Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind: Placebo (N=60) | Double Blind: JNJ-64565111 5.0 mg (N=59) | Double Blind: JNJ-64565111 7.4 mg (N=118) | Double Blind: JNJ-64565111 10.0 mg (N=118) | Open Label: Liraglutide 3.0 mg (N=119)
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 3 | 0 | 3 | 1
Abdominal Distension (Gastrointestinal disorders) | 2 | 4 | 6 | 6 | 7
Abdominal Pain (Gastrointestinal disorders) | 1 | 2 | 8 | 4 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 2 | 10 | 3 | 8
Constipation (Gastrointestinal disorders) | 3 | 7 | 20 | 21 | 20
Diarrhoea (Gastrointestinal disorders) | 3 | 8 | 24 | 23 | 27
Dry Mouth (Gastrointestinal disorders) | 1 | 4 | 6 | 5 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 5 | 18 | 13 | 9
Eructation (Gastrointestinal disorders) | 0 | 4 | 14 | 16 | 5
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 5 | 13 | 12 | 9
Nausea (Gastrointestinal disorders) | 4 | 30 | 80 | 79 | 48
Vomiting (Gastrointestinal disorders) | 0 | 12 | 47 | 64 | 20
Fatigue (General disorders) | 2 | 7 | 15 | 17 | 5
Injection Site Bruising (General disorders) | 4 | 2 | 1 | 2 | 1
Gastroenteritis (Infections and infestations) | 3 | 1 | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 9 | 5 | 11 | 6 | 10
Pharyngitis (Infections and infestations) | 3 | 0 | 2 | 0 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 0 | 4 | 2 | 6
Urinary Tract Infection (Infections and infestations) | 3 | 4 | 10 | 7 | 5
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 2 | 6 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 10 | 16 | 20 | 10
Dysgeusia (Nervous system disorders) | 1 | 4 | 3 | 2 | 0
Headache (Nervous system disorders) | 6 | 7 | 20 | 8 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT03486392/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT03486392/SAP_001.pdf